CLINICAL TRIAL: NCT00005623
Title: A Phase III, Randomized, Multicenter, Placebo-Controlled, Double-Blind Clinical Trial to Study the Efficacy and Safety of CyPat (Cyproterone Acetate [CA]) for the Treatment of Hot Flashes Following Surgical or Chemical Castration of Prostate Cancer Patients and Its Impact on the Quality of Life in These Patients
Brief Title: Cyproterone Acetate in Treating Hot Flashes Following Surgical or Chemical Castration for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barr Laboratories (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000067765; BARR-PCA-301
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2003-12

CONDITIONS: Hot Flashes; Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer; hot flashes
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Cyproterone Acetate

INTERVENTIONS:
Drug: cyproterone acetate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Cyproterone acetate may be effective treatment for hot flashes following surgical or chemical castration for prostate cancer. It is not yet known which regimen of cyproterone acetate is more effective for hot flashes.

PURPOSE: Randomized phase III trial to determine the effectiveness of cyproterone acetate in treating patients who have hot flashes following surgical or chemical castration for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of cyproterone acetate in patients with hot flashes following bilateral orchiectomy or medical castration for prostate cancer.
* Compare the effectiveness of two doses of cyproterone acetate in these patients.
* Determine the safety of this regimen in these patients.
* Determine the impact of this regimen on the quality of life of these patients.

OUTLINE: This is a randomized, double-blind, placebo controlled study.

Patients receive one of two doses of oral cyproterone acetate or placebo for 12 weeks, followed by a 6-9 month open label extension period with all patients receiving cyproterone acetate.

Quality of life is assessed.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prostate cancer patients who have undergone bilateral orchiectomy or medical castration (LHRH agonist drugs) and are experiencing hot flashes
* Hot flashes are defined as:

  * At least 3 to 4 moderate to severe hot flashes per day or 21 per week at baseline
  * Present at least 1 month prior to study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Greater than 12 months

Hematopoietic:

* WBC at least 3,000/uL
* Platelet count at least 75,000/uL
* Hemoglobin at least 6.2 mmol/L

Hepatic:

* Bilirubin no greater than 1.8 mg/dL
* SGPT no greater than 96 u/L
* SGOT no greater than 90 u/L
* LDH no greater than 600

Renal:

* BUN no greater than 42 mg/dL
* Creatinine no greater than 3.39 mg/dL

Cardiovascular:

* No cardiovascular risks (e.g., history of angina pectoris) unless controlled by medical or surgical therapy
* No known history of thromboembolic disease

Other:

* Comprehend and understand English language
* No other prior malignancy within the past 5 years except treated squamous or basal cell skin cancer or superficial bladder carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least a 4 week washout period is required if prior antineoplastic or cytotoxic chemotherapy has been used

Endocrine therapy:

* At least a 4 week washout period is required if prior estrogens, antiandrogens (e.g., flutamide or bicalutamide), progestational agents, or corticosteroids have been used
* No concurrent herbal medications with known hormonal ingredients (i.e., phytoestrogens)

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* At least a 4 week washout period is required if prior clonidine or monoamine oxidase inhibitors have been used

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Lewis, MD, Study Chair — MBCCOP - Medical College of Georgia Cancer Center
Locations (1):
- Barr Laboratories, Incorporated, Pomona, New York, United States